CLINICAL TRIAL: NCT06142136
Title: A Randomised Comparative Study of the Effect of LYL Love Your Life ® sunD3 LYL Micro™ Vitamin D Sublingual Spray on Vitamin D3 Levels in the Blood Compared to Other Forms of Vitamin D3 - Oral Oil Droplets and Capsules
Brief Title: The Effect of Vitamin D Sublingual Spray on Vitamin D3 Levels in the Blood Compared to Other Forms of Vitamin D3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 250321-6L
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2021-03

CONDITIONS: Vitamin D3 Deficiency
MeSH Terms: interventions — Capsules

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin D3 sublingual sprayable microemulsion. (Active Comparator): Total participants: 34 participants Duration: 30 days.
  Interventions: Dietary Supplement: Vitamin D substitution with sublingual sprayable microemulsion.
- Vitamin D3 oil droplets. (Active Comparator): Total participants: 33 participants Duration: 30 days.
  Interventions: Dietary Supplement: Vitamin D substitution with oil droplets
- Vitamin D3 capsules. (Active Comparator): Total participants: 32 participants Duration: 30 days.
  Interventions: Dietary Supplement: Vitamin D substitution with capsules

INTERVENTIONS:
Dietary Supplement: Vitamin D substitution with sublingual sprayable microemulsion. — Participants received sublingual sprayable microemulsion of vitamin D3 4000 IU daily for 30 days.
  Arms: Vitamin D3 sublingual sprayable microemulsion.
Dietary Supplement: Vitamin D substitution with oil droplets — Participants received oil droplets of vitamin D3 4000 IU daily for 30 days.
  Arms: Vitamin D3 oil droplets.
Dietary Supplement: Vitamin D substitution with capsules — Participants received capsules of vitamin D3 4000 IU daily for 30 days.
  Arms: Vitamin D3 capsules.

SUMMARY:
The randomized comparative study was performed on 99 outpatients with below 30 ng/ml of vitamin D. Participants were randomized into three groups to receive vitamin D3 supplementation in three different forms - sublingual spray, oral oil droplets, and capsules. Each participant received vitamin D3 4000 IU daily for 30 days and the vitamin D levels were measured before and after the intervention.

DETAILED DESCRIPTION:
This randomized comparative study was performed in Liepaja, Latvia, on 99 outpatients, with vitamin D levels below 30 ng/ml. Participants were randomized into three groups to receive vitamin D3 supplementation in three different forms - sublingual spray, oral oil droplets, and capsules. Before intervention blood samples were taken to determine vitamin D3 level, creatinine, and GFR, each participant received vitamin D3 4000 IU daily for 30 days. After that blood test was performed again, to measure changes in vitamin D3 levels in the blood. Participants answered the questionnaire to collect information about things that might affect vitamin D3 levels, such as dietary habits, physical activities, usage of sunscreen, compliance, etc.

ELIGIBILITY:
Inclusion Criteria:

* Vitamin D3 level in the blood below 30 ng/ml.

Exclusion Criteria:

* Celiac disease, Crohn's disease, ulcerative colitis, autoimmune gastritis.
* Patients with mental health problems.
* Vitamin D level ≥ 30 ng/ml.
* Pregnant women.
* Any other illness or condition that the researcher deemed may interfere with the results.
* Patients who refuse the studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-03-28 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Changes in vitamin D level in the blood depending on the received vitamin D form. | 30 days
  The study's primary outcome is to demonstrate the efficacy of sprayable microemulsion of cholecalciferol on the increase in circulating vitamin D levels over a period of 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Valdis Pirags, MD, PhD, Principal Investigator — Pauls Stradins Clinical University Hospital
Locations (1):
- Pauls Stradins Clinical Univeristy Hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No